CLINICAL TRIAL: NCT02156258
Title: Acquisition of Digital Mammography and Breast Images for Clinical Evaluation of FujifilmDigital Breast Tomosynthesis
Brief Title: Acquisition of Breast Mammography Images
Status: Completed | Type: Observational
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FMSU2013-004A
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Breast Cancer
Keywords: Imaging; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Diagnostic Cases: Collection of cases that were scheduled for biopsy (BI-RADS 4 or 5) using Full Field Digital Mammography (FFDM) Mammography and Digital Breast Tomosynthesis (DBT) Mammography
  Interventions: Device: FFDM Mammography; Device: DBT Mammography
- Recall Cases: Collection of Imaging Recall Cases (were scheduled for additional imaging due an assessment of BI-RADS 0) using FFDM Mammography and DBT Mammography
  Interventions: Device: FFDM Mammography; Device: DBT Mammography
- Screening Cases: Collection of cases who underwent routine screening mammography using FFDM Mammography and DBT Mammography
  Interventions: Device: FFDM Mammography; Device: DBT Mammography

INTERVENTIONS:
Device: FFDM Mammography — Standard mammography image collection
Device: DBT Mammography — Collection of breast images using DBT mammography

SUMMARY:
This is a case collection study of breast images using standard and new mammography technology.

DETAILED DESCRIPTION:
This image acquisition study is designed to acquire the study image data and establish and document the clinical findings for each subject. This study will create a library of image data that will be used for future projects.

ELIGIBILITY:
Inclusion Criteria:

For Screening Subjects

* Be at least 40 years of age, are
* Asymptomatic,
* Scheduled for a routine screening mammogram

For Recall Subjects

* Be at least 18 years of age,
* Received a BIRADS 0 within the last 60 days
* Are recalled for additional imaging

For Diagnostic Subjects

* Be at least 18 years of age,
* Scheduled for a biopsy due to an assessment of Breast Imaging and Reporting Data (BI-RADS®) 4 or 5 after diagnostic work-up of a suspicious screening or clinical finding within the last 60 days.
* Understand requirements and willing to participate in study

Exclusion Criteria:

* Presence of a breast implant.
* Women with only a single breast; for example, post mastectomy patients.
* Is pregnant or believes she may be pregnant.
* A woman who has delivered and who has expressed the intention to breast-feed or is currently breast-feeding.
* A woman who has significant existing breast trauma within the last one year.
* Have self-reported severe non-focal or bilateral breast pain affecting subject's ability to tolerate digital mammography and/or breast tomosynthesis examinations.
* A woman who has had a mammogram performed for the purpose of therapy portal planning within the last year.
* Cannot, for any known reason, undergo follow-up digital mammography and/or breast tomosynthesis examinations (where clinically indicated) at the participating institution.
* Is an inmate (see US Code of Federal Regulations 45CFR46.306).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of at least 200 cancer, 175 recall cases and 350 negative/benign cases will be accumulated
Sampling Method: Non-Probability Sample
Enrollment: 1232 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Etta D Pissano, MD, Principal Investigator — Medical University of South Carolina
Locations (5):
- United States (5):
  - Scottsdale Medical Imaging, Ltd, Scottsdale, Arizona
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Elizabeth Wende Breast Care, LLC, Rochester, New York
  - University of North Carolina - at Chapel Hill, Chapel Hill, North Carolina
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic Cases: Collection of diagnostic cases (scheduled for biopsy due to BI-RADS 4 or 5) using Full Field Digital Mammography (FFDM) Mammography and Digital Breast Tomosynthesis (DBT) Mammography
  FFDM Mammography: Standard mammography image collection
  DBT Mammography: Collection of breast images using DBT mammography
- Recall Cases: Collection of Imaging Recall Cases using FFDM Mammography and DBT Mammography
  FFDM Mammography: Standard mammography image collection
  DBT Mammography: Collection of breast images using DBT mammography
- Screening Cases: Collection of Screening Cases (underwent routine screening mammography) using FFDM Mammography and DBT Mammography
  FFDM Mammography: Standard mammography image collection
  DBT Mammography: Collection of breast images using DBT mammography
Period: Overall Study
Arm/Group | Diagnostic Cases | Recall Cases | Screening Cases
Started | 674 | 203 | 355
Completed | 642 | 124 | 244
Not Completed | 32 | 79 | 111

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diagnostic Cases | Recall Cases | Screening Cases | Total
Number analyzed (Participants) | 674 | 203 | 355 | 1232
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 518 | 164 | 274 | 956
  >=65 years | 156 | 39 | 81 | 276
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 674 | 203 | 355 | 1232
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 100 | 32 | 26 | 158
  Not Hispanic or Latino | 564 | 161 | 316 | 1041
  Unknown or Not Reported | 10 | 10 | 13 | 33
Region of Enrollment [Number; unit: participants]
  United States | 674 | 203 | 355 | 1232

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Whom Study Image Data Were Collected
Description: This study created a library of image data to be used in future projects, future product development and regulatory submissions. There was no analysis conducted aside from confirmation of complete images and collected data , as this was merely a collection of images to be used in future reader studies. Sites were provided a target distribution of diagnostic, recall and screening cases to obtain.
Time Frame: 20 Months
Population: Difference between enrolled and analyzed are those that were discontinued due to not returning for 1 year follow-up, etc. All cases were reviewed to ensure complete images and data, that was the extent of the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Cases | Recall Cases | Screening Cases
Number analyzed (Participants) | 674 | 203 | 355
Participants | 642 | 124 | 244

ADVERSE EVENTS:
Time Frame: 20 months
Description: Same definition applies for this study as indicated from clinicaltrials.gov.
Arm/Group | Diagnostic Cases | Recall Cases | Screening Cases
All-Cause Mortality (participants affected / at risk) | 0/674 | 0/203 | 0/355
Serious Adverse Events (participants affected / at risk) | 0/674 | 0/203 | 0/355
Other Adverse Events (participants affected / at risk) | 1/674 | 0/203 | 0/355
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diagnostic Cases (N=674) | Recall Cases (N=203) | Screening Cases (N=355)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — One subject fainted during the mammogram. The enrolling center determined that the event was not related to the study procedure and not related to the investigational device. The subject fully recovered before leaving the center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No